CLINICAL TRIAL: NCT07321964
Title: The Effect of MediYoga on Quality of Life, Blood Pressure and Heart Rate Among Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: The Effect of a Digital MediYoga Program on Quality of Life, Blood Pressure and Heart Rate Among Patients With Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Sophiahemmet (Unknown)
Responsible Party: Principal Investigator, Signe Stelling Risom, Associate Professor, PhD, RN, Senior Researcher, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-24084633
Record Dates: First submitted 2025-09-26; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation (Paroxysmal); Quality of Life; Mental Health
Keywords: Digital Health Intervention; Atrial Fibrillation; Yoga; Quality of Life; Nursing
MeSH Terms: conditions — Atrial Fibrillation; Psychological Well-Being | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group I, yoga 20 minutes x3 pr week (Experimental)
  Interventions: Behavioral: Yoga 20 minutes
- Intervention group II, yoga 60 minutes x1 pr week (Experimental)
  Interventions: Behavioral: Yoga 60 minutes
- Control group (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Yoga 20 minutes — The intervention consists of 60 minutes of weekly MediYoga over a 12-week period. Participants in the intervention group may choose whether they prefer to practice yoga for 20 minutes three times per week, or for 60 minutes once per week. The yoga sessions are delivered via a smartphone application, guiding participants through the sessions with both video and audio. In addition, participants are required to complete three questionnaires and measure blood pressure and heart rate at baseline, and at 3 and 6 months of follow-up.
  Other Names: MediYoga; MOSI
  Arms: Intervention Group I, yoga 20 minutes x3 pr week
Behavioral: Yoga 60 minutes — The intervention consists of 60 minutes of weekly MediYoga over a 12-week period. Participants in the intervention group may choose whether they prefer to practice yoga for 20 minutes three times per week, or for 60 minutes once per week. The yoga sessions are delivered via a smartphone application, guiding participants through the sessions with both video and audio. In addition, participants are required to complete three questionnaires and measure blood pressure and heart rate at baseline, and at 3 and 6 months of follow-up.
  Other Names: MediYoga; MOSI
  Arms: Intervention group II, yoga 60 minutes x1 pr week

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrythmia, associated with increased risk of stroke, heart failure, reduced quality of life (QoL), and psychological distress. This randomized controlled trial investigates the effect of MediYoga - a program incorporating deep breathing, low-intensity yoga, and meditation- on disease-specific QoL, blood pressure, and heart rate in 456 patients with paroxysmal AF. With a strong focus on sustainability, the study is fully digital: participants are recruited online, and the 12-week intervention is delivered through an application to smartphone. Additionally, the participants receive online support via Teams. Data will be collected at baseline, 3, 6, and 12 months. The primary outcome is disease specific QoL; secondary outcomes include blood pressure, heart rate, generic QoL, and psychological wellbeing.

Qualitative interviews will explore patients' experiences with the intervention.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac arrythmia, affecting approximately 3% of the adult population. AF is associated with substantial morbidity including increased risk of stroke and heart failure, and increased mortality risk. The risk of developing AF raises with age hence the prevalence of AF is expected to increase substantially in the future, due to increased average life expectancy. The costs from diagnostics, treatments, and in- and out-patient care, is likewise estimated to increase, because of the expanding proportion of old-er individuals, development of treatment options, and intensifying search for undiagnosed AF. Risk factors such as hypertension, coronary artery disease, obesity, type 2 diabetes, stress, alcohol overconsumption, smoking, and sleep apnea are also increasing in prevalence and are potent contributors to the development and progression of AF.

Various symptoms can occur during an AF episode, including dizziness, heart palpitations, chest pain, and fatigue. Standard treatment of AF include rhythm- and/or rate-control medications, electrical cardioversion, and in some cases catheter ablation. The treatment focuses on re-ducing symptoms and improving quality of life (QoL).

AF episodes can have negative impact on patient's physical and mental health, as well as so-cial life. Individuals with AF often report poorer QoL, and experience symptoms of stress, depression, and anxiety. Guidelines recommend self-care programs that reduce symptoms and enhance QoL and recommends regularly physical activity to improve overall cardiovascular health. Yoga has been shown to improve health-related quality of life (HRQoL), reduce blood pressure and heart rate, and reduce AF episodes in small studies in-cluding individuals with paroxysmal AF. MediYoga originates from Kundalini Yoga, and is based on deep breathing, combined with slow movements, meditation, and relaxation exercises. MediYoga is designed so that many of the exercises can be performed while seated.

The increasing proportion of older individuals living with AF, demands new ways of organizing and implement rehabilitation for patients. Tele-health, defined as the delivery of health-related services through digital communication technologies is eligible to provide yoga classes at home. Online interventions might increase the likelihood that participants complete the program, as it can be done in their own surroundings without required transportation. Remote recruitment has increasing potential, as it enhances the possibility to include participants from rural districts, who might not participate in onsite rehabilitation, due to the long distance to a rehabilitation center.

To our knowledge, this study is the first study to investigate the effect of an online yoga intervention for patients with symptomatic paroxysmal AF, using a complete online recruitment and implementation strategy.

This study is designed as a randomized controlled digital trial, and will be conducted as an international study with recruitment in both Denmark and Sweden. This study will be conducted as a parallel study with the Swedish study. No data will be transferred. The analyzes will be done separately but published in the same publication with comparisons between countries.

The study is designed as a three arm, randomized superiority trial. Participants will be randomly assigned to one of two groups (1:1) (I) control group including treatment as usual (TAU) alone, or (II) intervention group, in which participants will be allocated to one of two groups, based on their personal preferences; (IIa) performing yoga three times a week for 20 min or (IIb) performing yoga once a week for 60 minutes, for at total of 12 weeks, in addition to TAU

To explore how participants experience being a part of the study, 12-15 patients from each intervention group will be interviewed using qualitative methods. A semi-structured interview guide will be developed through the intervention period, as interesting themes arises. Questions will be formulated to both capture patients experience of the recruitment process and being a part of a study using health technology and remote participation, as well as how the patients experience carrying out the intervention using an app and being in their home. Data will be analyzed using thematic analysis.

All data are self-reported by participants; therefore, access to patient records is not required.

The primary outcome is the disease-specific questionnaire, ASTA. The validated form is divided into three parts: evaluation of the most recent episode of arrythmia and current medication assessment of symptom burden, including a 9-point symptom scale (ASTA symp-tom scale) with a 4-point response scale, and assessment of the HRQoL using a 13-point scale (ASTA scale) with the same 4-point response scale as the symptom scale. The ASTA scale is further divided into a physical and a mental subscale. Scores range from 0 to 100, with higher scores reflecting a higher symptom burden and a worse impact on HRQoL due to arrythmia.

The SF-36 is a standardized, validated, and reliable general HRQoL questionnaire containing 36 items.The items are divided into eight domains and two component summary scales reflecting physical and mental health re-spectively. The two summary scales are analysed on a 0-100 scale, where 100 represents the best possible HRQoL.

HADS is a reliable and validated instrument for screening for clinically relevant symptoms of anxiety and depression in patients. The scale consists of 14 items assessing how patients felt during the previous week. Patients must answer every question in a 4-point Likert scale from 0 to 3. Seven of the items assess the level of depression, and the remaining seven the level of anxiety. Scores are summarized separately for anxiety and depression, resulting in two scores with a range of 0-21. Higher scores indicate more symptoms of anxiety and depression.

In addition to the self-administrated questionnaires, Participants in both the intervention and control groups will be asked to measure their blood pressure and heart rate using a device provided by the research team. They will receive a detailed guide on how to perform these measurements at home, in accordance with the European Guidelines for the Management of Elevated Blood Pressure and Hypertension. Participants will be instructed to take their measurements in the morning, prior to breakfast and any medication intake. Additionally, they will be asked to empty their bladder, refrain from smoking for at least 30 minutes beforehand, and rest for 1-5 minutes before beginning. Blood pressure and heart rate should be measured three times, with 1-2 minutes between each reading. Participants will complete questionnaires and perform blood pressure and heart rate measurements at baseline, 3 and 6 months follow-up.

Sociodemographic characteristics including age, sex, occupational status, educational level, marital status, medication, and comorbidities will be collected via self-report at baseline.

Statistical Analysis Comparisons between the intervention and control groups will be made using Chi-square tests for proportions and repeated measures ANOVA for analyzing questionnaires, blood pressure, and heart rate. Student's t-test will be used for within-group anal-yses. Analysis of covariance (ANCOVA) will be used if a statistically significant relationship is shown between groups regarding demographic data. Drop-out rate will be registered in a flowchart and both per protocol and intent-to-treat analyses will be performed. The level of significance is set at p<0.05. The analysis will be performed by a blinded statistician.

If the intervention proves effective, the findings could contribute to a scalable, evidence-based model for remote AF rehabilitation, supporting the broader movement toward digital and patient-centered care in cardiology.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Diagnosed with paroxysmal atrial fibrillation
* EHRA score at 2 or more
* Owner of a smartphone or tablet
* Speaking and reading Danish
* No comorbidity that restricts them from participating in the intervention

Exclusion Criteria:

* Elevated TSH Hormone
* Participated in mindfulness or yoga exercise regularly at any point during the last two years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Arrythmia-Specific Symptoms and Health-Related Quality | Baseline, and at 3 and 6 months after enrollment
  The validated form is divided into three parts: (1) evaluation of the most recent episode of arrythmia and current medication (2) assessment of symptom burden, including a 9-point symptom scale (ASTA symptom scale) with a 4-point response scale, and (3) assessment of the HRQoL using a 13-point scale (ASTA scale) with the same 4-point response scale as the symptom scale. The ASTA scale is further divided into a physical and a mental subscale. Scores range from 0 to 100, with higher scores reflecting a higher symptom burden and a worse impact on HRQoL due to arrythmia

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline, and at 3 and 6 months after enrollment
  The SF-36 is a standardized, validated, and reliable general HRQoL questionnaire containing 36 items. The questionnaire is commonly used in AF studies. The items are divided into eight domains and two component summary scales reflecting physical and mental health re-spectively. The two summary scales are analysed on a 0-100 scale, where 100 represents the best possible HRQoL.
Mental health | Baseline, and at 3 and 6 months after enrollment
  HADS is a reliable and validated instrument for screening for clinically relevant symptoms of anxiety and depression in patients. The scale consists of 14 items assessing how patients felt during the previous week. Patients must answer every question in a 4-point Likert scale from 0 to 3. Seven of the items assess the level of depression, and the remaining seven the level of anxiety. Scores are summarized separately for anxiety and depression, resulting in two scores with a range of 0-21. Higher scores indicate more symptoms of anxiety and depression
Blood pressure | Baseline, and at 3 and 6 months after enrollment
  Blood pressure
Pulse | At baseline, and 3 and 6 months after enrollment
  Pulse monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request
Supporting Information: Study Protocol, ICF